CLINICAL TRIAL: NCT04470921
Title: STOP OVarian CAncer; Implementation of the Opportunistic Salpingectomy in the Netherlands
Acronym: STOPOVCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1; 11515
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Risk Reduction; Ovarian Cancer
Keywords: Ovarian cancer; Opportunistic Salpingectomy; Prevention; Female sterilization; Risk reduction; Implementation
MeSH Terms: conditions — Risk Reduction Behavior; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Choice for Opportunistic Salpingectomy: Women who will undergo a gynaecological surgery in which currently both ovaries and fallopian tubes would be preserved, can opt for an opportunistic salpingectomy.
  Interventions: Procedure: Opportunistic Salpingectomy

INTERVENTIONS:
Procedure: Opportunistic Salpingectomy — An opportunistic salpingectomy refers to removal of the fallopian tubes without the ovaries during (laparoscopic) interventions for benign (gynaecological) disease to reduce the number of ovarian cancer cases.

SUMMARY:
The aim of this study is to optimize implementation of the opportunistic salpingectomy throughout the Netherlands.

DETAILED DESCRIPTION:
The investigators aim to optimize implementation of opportunistic salpingectomy throughout the Netherlands. The investigators will evaluate the implementation by enrolling patients in a database to evaluate healthcare experiences and to register EOC diagnosis and vital status through yearly PALGA (the nationwide network and registry of histopathology and cytopathology in the Netherlands) and municipal administration searches. In addition, the investigators will perform medical record check to assess which percentage of eligible women have been offered OS.

The investigators expect that a decision aid will be a necessary tool for the decision whether women opt for an OS or not, based on their personal values. After development of the tool(s), the investigators will evaluate the implementation process.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 years
* Undergoing gynaecological surgery in which currently both ovaries and fallopian tubes would be preserved
* Childbearing completed
* Able to understand the written or spoken Dutch language
* Consent for enrolment in database
* Consent for yearly checks of PALGA database and municipal administration

Exclusion Criteria:

* Age under 30 years
* Undergoing surgery without residual ovarian tissue
* Child wish
* Unable to understand the written or spoken Dutch language
* Previous bilateral salpingectomy
* Previous bilateral salpingo-oophorectomy

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who will undergo a gynaecological surgery in which currently both ovaries and fallopian tubes would be preserved, can opt for an opportunistic salpingectomy.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Offered Opportunistic Salpingectomy (OS) | 2019 - 2023
  Number of eligible women who have actually been offered an opportunistic salpingectomy in the Netherlands.
Implementation effect of Opportunistic Salpingectomy (OS) | 2019-2023
  The effect of our implementation efforts on the number of eligible women who have actually been offered an opportunistic salpingectomy in the Netherlands.

SECONDARY OUTCOMES:
Influencing factors implementation Opportunistic Salpingectomy (OS) | 2019-2020
  Determine factors that impede and facilitate nationwide implementation of Opportunistic Salpingectomy.
Implementation tools | 2019-2020
  Implementation tools, developed based on the barriers and facilitators of the influencing factors.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne A de Hullu, MD, PhD, Principal Investigator — University Medical Center Nijmegen; Jurgen MJ Piek, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Rosella PM Hermens, PhD, Principal Investigator — Scietific Institute for Quality of Healthcare, UMC Nijmegen
Locations (27):
- Netherlands (27):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - OLVG, Amsterdam
  - Academic Medical Centrum, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia hospital, Breda
  - Reinier de Graaf, Delft
  - Slingeland Hospital, Doetinchem
  - Albert Schweitzer hospital, Dordrecht
  - Catharina Hospital, Eindhoven
  - Medical Spectrum Twente, Enschede
  - Martini hospital, Groningen
  - Spaarne Gasthuis, Haarlem
  - Ziekenhuisgroep Twente, Hengelo
  - Medical Center Leewarden, Leeuwarden
  - Leids University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - St Antonius, Nieuwegein
  - Radboud UMC, Nijmegen
  - Canisius Wilhelmina Hospital, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medical Center Westeinde, The Hague
  - Elisabeth-Tweesteden Hospital, Tilburg
  - Diakonessenhuis, Utrecht
  - Maxima Medical Center, Veldhoven
  - VieCuri Medical Center, Venlo
  - Sint Jans Gasthuis, Weert
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoon SH, Kim SN, Shim SH, Kang SB, Lee SJ. Bilateral salpingectomy can reduce the risk of ovarian cancer in the general population: A meta-analysis. Eur J Cancer. 2016 Mar;55:38-46. doi: 10.1016/j.ejca.2015.12.003. Epub 2016 Jan 8. PMID 26773418
- [Background] Kwon JS, McAlpine JN, Hanley GE, Finlayson SJ, Cohen T, Miller DM, Gilks CB, Huntsman DG. Costs and benefits of opportunistic salpingectomy as an ovarian cancer prevention strategy. Obstet Gynecol. 2015 Feb;125(2):338-345. doi: 10.1097/AOG.0000000000000630. PMID 25568991
- [Background] van Lieshout LAM, Steenbeek MP, De Hullu JA, Vos MC, Houterman S, Wilkinson J, Piek JM. Hysterectomy with opportunistic salpingectomy versus hysterectomy alone. Cochrane Database Syst Rev. 2019 Aug 28;8(8):CD012858. doi: 10.1002/14651858.CD012858.pub2. PMID 31456223
- [Background] Steenbeek MP, van Lieshout LAM, Aarts JWM, Piek JMJ, Coppus SFPJ, Massuger LFAG, Hermens RPMG, de Hullu JA. Factors influencing decision-making around opportunistic salpingectomy: a nationwide survey. J Gynecol Oncol. 2019 Jan;30(1):e2. doi: 10.3802/jgo.2019.30.e2. Epub 2018 Apr 30. PMID 30479086
- [Background] Committee opinion no. 620: Salpingectomy for ovarian cancer prevention. Obstet Gynecol. 2015 Jan;125(1):279-281. doi: 10.1097/01.AOG.0000459871.88564.09. PMID 25560145
- [Background] Salvador S, Scott S, Francis JA, Agrawal A, Giede C. No. 344-Opportunistic Salpingectomy and Other Methods of Risk Reduction for Ovarian/Fallopian Tube/Peritoneal Cancer in the General Population. J Obstet Gynaecol Can. 2017 Jun;39(6):480-493. doi: 10.1016/j.jogc.2016.12.005. PMID 28527613